CLINICAL TRIAL: NCT06306183
Title: Does Vitamin C Provide an Analgesic Effect on Acute Musculoskeletal Injury After an Emergency Department Visit: A Double-Blind Randomized Control Trial
Brief Title: Effect of Vitamin C on Pain Reduction After an Emergency Department Visit
Acronym: Vicamed
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Hopital de l'Enfant-Jesus (Other); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Raoul Daoust, Dr Emergency Medicine, Professor, Clinician Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-2829
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Pain, Acute
Keywords: Vitamin C; NSAID; Emergency department; Pain; RCT
MeSH Terms: conditions — Acute Pain; Emergencies; Pain | interventions — Acetaminophen; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen and Vitamin C with Naproxen rescue (Experimental): 900 mg vitamin C taken orally twice a day Extended-release acetaminophen 650 mg two pills every eight hours regularly
  Naproxen 500 mg as a rescue medication
  Interventions: Dietary Supplement: Acetaminophen and Vitamin C with Naproxen rescue
- Acetaminophen and Placebo with Naproxen rescue (Placebo Comparator): Placebo taken orally twice a day Extended-release acetaminophen 650 mg two pills every eight hours regularly
  Naproxen 500 mg as a rescue medication

INTERVENTIONS:
Dietary Supplement: Acetaminophen and Vitamin C with Naproxen rescue — 900 mg vitamin C taken orally twice a day (one in the morning and one in the evening) for a 7-day period after ED discharge for the treatment arm used in combination with extended-release acetaminophen 650 mg two pills every eight hours regularly.
  Naproxen 500mg as rescue medication if still in pain 60 minutes after treatment with acetaminophen.
  Arms: Acetaminophen and Vitamin C with Naproxen rescue
Other: Acetaminophen and Placebo with Naproxen rescue — Placebo taken orally twice a day (one in the morning and one in the evening) for a 7-day period after ED discharge for the treatment arm used in combination with extended-release acetaminophen 650 mg two pills every eight hours regularly.
  Naproxen 500mg as rescue medication if still in pain 60 minutes after treatment with acetaminophen.

SUMMARY:
Emergency department (ED) clinicians often prescribe anti-inflammatory drugs (NSAIDs) to manage acute musculoskeletal (MSK) pain (e.g.: fracture, sprain, back pain). However, even short-term NSAIDs use can have significant gastrointestinal, cardiovascular, MSK and renal adverse effects. For this reason, some patients cannot take or tolerate NSAIDs. Recent evidence has shown that vitamin C has some analgesic and anti-inflammatory properties particularly in postoperative context and prevent specific types of chronic pain. Furthermore, vitamin C is safe and associated with very few adverse events. The primary objective of this study is to determine whether vitamin C can reduce pain intensity during a seven-day period following an ED visit for acute MSK pain.

The investigators propose to compare two groups of patients, one receiving 900 mg of vitamin C to another receiving a placebo, twice a day for seven days. Both groups will consume acetaminophen slow release 650 mg two pills every eight hours regularly. Naproxen 500 mg (NSAID) will be used as a rescue medication if the patient's pain is not relieved. Participants will be ≥18 years of age, treated in ED for acute MSK pain present for less than 48 hours with pain intensity at triage of ≥ 4 on a 0-10 numeric rating scale, and discharged by an ED clinician with an NSAIDs prescription without opioids. The level of pain intensity during a seven-day period will be assessed daily using an electronic or paper diary, as well as pain relief, pain medication consumption, and adverse events. Three months after the injury, participants will also be contacted to assess the presence of chronic pain. The investigators hypothesized that vitamin C will reduce pain intensity and chronic pain development at three months.

This research could provide a safe alternative to patients who are unable to take NSAIDs. It may also contribute to the reduction of the burden associated with chronic pain development.

DETAILED DESCRIPTION:
Background and Importance: Nonsteroidal anti-inflammatory drugs (NSAIDs) have proven their efficacy and compared advantageously to opioids in treating acute musculoskeletal (MSK) pain. However, even short-term NSAIDs use for acute pain management after an emergency department (ED) discharge can have significant gastrointestinal, cardiovascular, musculoskeletal and renal adverse effects. Recent evidence has shown that vitamin C has, in addition to its antioxidant effect, some analgesic and anti-inflammatory properties. Its analgesic effect has been explored mostly in short-term postoperative context or in disease-specific chronic pain prevention, but never after acute pain from MSK injuries, which are often seen in EDs.

Goal(s) / Research Aims: The primary aim is to evaluate the effectiveness of vitamin C in reducing pain intensity during a seven-day period following ED discharge for an acute MSK pain complaint. The secondary aims are to compare both treatment groups for rescue medication use, average pain relief and adverse events during a seven-day follow-up, and at three months for chronic pain incidence.

Methods / Approaches / Expertise: The investigators will conduct a pragmatic five-center, double-blind randomized placebo-controlled trial (RCT) with 546 participants equally distributed in two arms; one group receiving 900 mg of vitamin C and another one receiving a placebo, twice a day for seven days. Both groups will consume acetaminophen slow release 650 mg two pills every eight hours regularly. Naproxen 500 mg will be used as a rescue medication if the patient's pain is not relieved more than one hour after acetaminophen consumption. Participants will be aged ≥18 years, treated in the emergency department for acute MSK injury present for less than 48 hours with a pain intensity at triage of ≥ 4 on a numerical rating scale (NRS) of 0-10, and scheduled for discharge by an emergency clinician with an NSAIDs prescription without opioids. Daily pain intensity during the seven-day period will be assessed via a previously tested electronic or paper diary. In addition, patients will report their daily rescue pain medication use, pain relief, and adverse events. Three months after the ED visit, participants will be contacted to evaluate chronic pain development.

The investigators hypothesized that vitamin C will reduce pain intensity during a seven-day follow-up for ED discharged patients treated for acute MSK pain. This project brings together a committed, multidisciplinary research team composed of five study sites having previously collaborated on large multicenter RCT studies. All required instruments have been successfully used during an ongoing Canadian Institutes of Health Research (CIHR) grant, a non-objection letter from Health Canada has been already requested and the investigators have secured a provider for both study drugs, all this ensuring a rapid study implementation.

Expected Outcomes: The investigators will provide the following outcomes for patients receiving vitamin C and placebo: pain intensity, rescue medication use, pain relief, and side effects for one-week post-discharge and chronic pain incidence at three months. Confirmation of the vitamin C analgesic effect for acute MSK pain could help patients who are unable to consume or are at risk of complications from NSAIDS. It may also contribute to the reduction of the burden associated with chronic pain development.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Treated in the ED for acute MSK pain present ≤ 48 hours at triage (time to presentation for most acute MSK pain in our previous study)
3. Numerical rating scale (NRS) pain intensity at triage of ≥ 4 on a 0-10 scale
4. Discharged with instructions to take an NSAID for pain (need determined by treating clinicians)
5. French or English-speaking

Exclusion Criteria:

1. Received an opioid prescription at ED discharge
2. Currently using vitamin C supplements
3. Active cancer
4. Currently treated for chronic pain
5. Unable to fill out a diary or unavailable for follow-up
6. Allergy, to milk (lactose in the placebo), vitamin C, acetaminophen or NSAIDs
7. Treated with cyclosporine or warfarin (interaction with vitamin C)
8. Pre-existing oxalate nephropathy, liver cirrhosis or hemochromatosis
9. Pregnant ≥ 20 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender is self identified by participants.
Enrollment: 546 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Daily pain intensity | Seven days
  The daily pain intensity will be measured with validated a 0-100 plasticized visual analog scale (VASp) provided to participants during the initial ED visit and documented in the electronic or paper diary.

SECONDARY OUTCOMES:
NSAIDs consumption | Seven days
  Consumption of NSAIDs rescue medication after seven days. Numbered in seven-day diary and counted at the one-week questionnaire.
Pain relief | Seven days
  Participants will be asked each day during the seven-day follow-up if their pain has been adequately relieved during the day (yes or no). This will be reported as a percentage.
New analgesic prescriptions | Seven days
  Numbered and of new pain medication prescription received during follow-up, even opioids.
Adverse events | Seven days
  We will document during the one-week questionnaire if any of the following adverse events were experienced during the seven-day period: nausea, vomiting, constipation, dizziness, drowsiness, sweating, weakness, or other adverse events.
Quality of life improvement at seven days | Seven days
  Quality of life will be evaluated during the one-week interview with the validated 12-Item Short Form Survey (SF-12 questionnaire). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Quantity of Healthcare visits | Seven days
  Participants will be asked about the number of all unscheduled or scheduled healthcare visits related to their initial pain condition during the 1-week questionnaire.
Prevalence of chronic pain | 90 days
  Questionnaire at 90 days. Chronic pain will be defined as pain intensity of ≥ 4 on the NRS (0-10) persistent or that reoccurs on most days after three months.
Prevalence of complex regional pain syndromes for limb fractures | 90 days
  For participants with limb fractures who are still in pain at 90 days, an in-person visit will be scheduled to evaluate the presence of complex regional pain syndrome as defined by the Budapest criteria, which includes a physical examination.
  To make the clinical diagnosis, the following criteria must be met:
  Continuing pain, which is disproportionate to any inciting event.
  Must report at least one symptom in all four of the following categories:
  Sensory Vasomotor Sudomotor/oedema Motor/trophic
  Must display at least one sign at time of evaluation in two or more of the following categories:
  Sensory Vasomotor Sudomotor/oedema Motor/trophic
  There is no other diagnosis that better explains the signs and symptoms.
Quality of life improvement at 90 days | 90 days
  Quality of life will be evaluated during the three-month interview with the validated 12-Item Short Form Survey (SF-12 questionnaire). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Daoust, MD MSc, Principal Investigator — Université de Montréal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada